CLINICAL TRIAL: NCT06891365
Title: Investigation of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of NNC0581-0001 in Participants With Hepatic Steatosis and Suspected Steatohepatitis
Brief Title: Multiple Dose Study for a New Medication to Potentially Treat Liver Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6581-4981; U1111-1298-9628 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers; Hepatic Steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: NNC0581-0001 (Dose 1) (Experimental): Participants will receive a subcutaneous (s.c) injection of either NNC0581-0001 Dose 1 or a matching placebo once monthly.
  Interventions: Drug: NNC0581-0001; Drug: Placebo (NNC0581-0001)
- Cohort 2: NNC0581-0001 (Dose 2) (Experimental): Participants will receive a s.c injection of either NNC0581-0001 Dose 2 or a matching placebo once monthly.
  Interventions: Drug: NNC0581-0001; Drug: Placebo (NNC0581-0001)

INTERVENTIONS:
Drug: NNC0581-0001 — NNC0581-0001 will be administered subcutaneously.
Drug: Placebo (NNC0581-0001) — Placebo matched to NNC0581-0001 will be administered subcutaneously.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of NNC0581-0001 in participants with hepatic steatosis and suspected steatohepatitis (increased liver fat and suspected inflammation). NNC0581-0001 will be given in 2 different dose levels as injection under the skin (once per month for 3 months). Participants will either get NNC0581-001 or Placebo (dummy treatment). Which treatment participants get is decided by chance. NNC0581-0001 is a new medicine which cannot be prescribed by doctors. The study will last about 58 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* Male or female (of non-childbearing potential) aged 18-64 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) 25.0 to 39.9 kilogram per square meter (kg/m^2) (both inclusive) at screening.
* Liver fat content measured by magnetic resonance imaging - estimated proton density fat fraction (MRI-PDFF) greater than or equal to (>=) 10 percent and liver stiffness greater than 8 kilopascal (kPa) as measured by FibroScan® (vibration-controlled transient elastography [VCTE™]).

Additional inclusion criteria for participants in the open-label liver biopsy cohort apply:

* Alanine aminotransferase (ALT) in men greater than (>) 30 units per liter (U/L), women > 19 U/L
* Liverstiffness, measured by FibroScan® (VCTE) > 8 kPa and less than (<) 12 kPa
* Informed consent obtained at screening for a liver biopsy to be performed at baseline and post-treatment.

Note: Participants with confirmed metabolic dysfunction-associated steatohepatitis (MASH), based on a prior liver biopsy, can be included in the open-label cohort.

Exclusion Criteria:

* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Any laboratory safety parameter, at screening, outside the extended laboratory ranges, and considered clinically significant per the principal investigator (see laboratory provided reference ranges for specific values). Of note, re-screening or re-sampling is NOT allowed if the individual has failed one of the exclusion criteria related to the following laboratory parameters:
* ALT >= 3 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) >= 3 × ULN
* Bilirubin > 1.5 × ULN
* Estimated glomerular filtration rate (eGFR) < 60 milliliter per minute per 1.73 square meters (mL/min/1.73 m^2) at screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From 1st dose (day 1) until completion of the end of study visit at week 52
  Measured as count of events.

SECONDARY OUTCOMES:
AUC0-32h: The area under the NNC0581-0001 plasma concentration-time curve from time zero to 32 hours after each of the three doses | From dosing (day 1 in each treatment period) to 32 hours post dose
  Measured in nanogram hour per mililitre (ng*h/mL).
Cmax: The maximum concentration of NNC0581-0001 in plasma after each dose of three doses | From dosing (day 1 in each treatment period) to 32 hours post dose
  Measured in nanogram per mililitre(ng/mL).
Tmax: The time from dose administration to maximum plasma concentration of NNC0581-0001 after each dose of three doses | From dosing (day 1 in each treatment period) to 32 hours post dose
  Measured in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Parexel CPRU, Level 7, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com